CLINICAL TRIAL: NCT03811093
Title: Comparing the Efficacy of a Dual-Frequency Laser-Emitting Device, the "Invisared-RED Elite", With a Sham Device as Therapy for the Loss of Adipose Tissue (Body Fat) and Aesthetics in Overweight Individuals
Brief Title: Comparing the Efficacy of a Dual-Frequency LLLT Device With a Sham Device as a Therapy for Adipose Tissue Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IR Technology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: invisa-RED_Trial
Record Dates: First submitted 2019-01-16; First posted 2019-01-22 (Actual); Results first posted 2019-06-04 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Body Weight; Fat Burn; Cellulite; Abdominal Fat; Adipose Tissue Atrophy
Keywords: Adipose, Fat, Aesthetics, Skin, Weight Reduction,
MeSH Terms: conditions — Obesity; Body Weight; Cellulite; Platelet Glycoprotein IV Deficiency; Weight Loss

STUDY DESIGN:
Intervention Model Description: The trial compared results between two groups of participants; the first group was treated using a fully functional device. The second, a control group, was treated utilizing a nonfunctional device. At the conclusion of nine (9) therapy sessions; the change in body fat percentage, the change in body fat in pounds, and inches lost of the two groups will be statistically analyzed to determine the efficacy of the invisa-RED Technology Elite as a weight loss therapy. Any medical errors will be included in the statistical analysis.
Who Masked: Participant, Care Provider
Masking Description: The trial will be conducted employing a double blind study methodology; participants will be randomly assigned to each group through a drawing, neither participants nor clinicians will know to which trial group they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Care as Usual Group (Experimental): A randomly selected group of 20 participants who received treatment per the prescribed trial protocol using a fully functional invisa-RED Technology Elite device. Treatment protocol was as follows: Participants will undergo nine (9) therapy sessions of 20 minutes each over a three week period; using a singular LLLT protocol setting for pulse (3.5s) and delay (0.2s), however power settings will be based on the participants Fitzpatrick Scale skin type. For skin types i and ii a power setting of 7 will be used, for skin types iii and iv a power setting of 6, for skin types v and vi a power setting of 4 will be employed.
  Interventions: Device: Care as Usual Group
- Sham Group (Placebo Comparator): A randomly selected group of 20 participants who will receive treatment per the prescribed trial protocol using a non functional invisa-RED Technology Elite device. (The sham device will be disabled and will deliver no low laser light energy during therapy.) Treatment protocol is as follows: Participants will undergo nine (9) therapy sessions of 20 minutes each over a three week period; using a singular protocol setting for pulse (3.5s) and delay (0.2s), however power settings will be based on the participants Fitzpatrick Scale skin type. For skin types i and ii a power setting of 7 will be used, for skin types iii and iv a power setting of 6, for skin types v and vi a power setting of 4 will be employed.
  Interventions: Device: Sham Group

INTERVENTIONS:
Device: Care as Usual Group — Each participant randomly assigned to the "Care As Usual Group" will undergo nine therapy sessions over three weeks using a fully functioning invisa-RED Technology Elite device.
  Arms: Care as Usual Group
Device: Sham Group — Each participant randomly assigned to the "Sham Group" will undergo nine therapy sessions over three weeks using a non functioning invisa-RED Technology Elite device.
  Arms: Sham Group

SUMMARY:
The trial was designed to provide empirical evidence with which to compare the efficacy and safety of the invisa-RED Technology Elite Low-level Laser Therapy (LLLT) device with a sham device as a placebo, when both are used in the treatment of individuals to reduce body fat and improve body aesthetics. At the conclusion of the trial; the change in body fat percentage, the change in total body fat in pounds, and total inches lost of the two groups were statistically analyzed to determine the efficacy of the invisa-RED Technology Elite when used for body fat (adipose tissue) loss and/or aesthetics therapy.

DETAILED DESCRIPTION:
The trial was designed to prove the efficacy and safety of the invisa-RED Technology Elite Low-level Laser Therapy (LLLT) device. The trial compared results between two groups; the first group was treated using a fully functional invisa-RED Technology Elite device; this group was designated the Usual Care Group.

The second, a control group, was treated utilizing a nonfunctional invisa-RED Technology Elite device; this group is referred to as the Sham Group.The sham device consisted of an invisa-RED Technology Elite device that will appear to operate as the Usual Care Group device to the operator and participants, but the laser diodes will be disabled and will receive no power providing a placebo effect. If staff or a participant questions the efficacy of the sham device, an assertion may be made that only a near infrared, non-visible frequency of light, is being employed.

The trial was conducted employing a double blind study methodology; participants were randomly assigned to each group through a drawing, neither participants nor clinicians knew to which trial group they were assigned. To ensure the double blind; treatment for the two groups occurred separately using clinicians exclusive to each group.

A simplified weight loss protocol was employed based on the "Consultation Protocol" from the invisa-Red Training Manual. All study participants received nine (9) therapy sessions of 20 minutes each; power settings were based on the participants Fitzpatrick Scale skin type. For skin types i and ii a power setting of 7 was used, for skin types iii and iv a power setting of 6, for skin types v and vi a power setting of 4 was employed. At the conclusion of the nine (9) therapy sessions; the change in weight of body fat, body fat as a percentage of total body weight, and inches lost of the two groups were statistically analyzed to determine the efficacy of the invisa-RED Technology Elite as a therapy to reduce adipose tissue. The occurrence of any medical errors were documented and included in the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

Any healthy individual.

Exclusion Criteria:

* If you are pregnant, trying to get pregnant or nursing laser light therapy should be received only after the end of these conditions. There is no evidence of harm to a an unborn baby however there have been no safety tests either, so for medical legal reasons we recommend never treating areas directly over a developing child.
* Individuals with hypertension, light sensitive epilepsy, cancer, heart disease, infectious skin disease, and severe varicose veins should not use this device.
* People suffering from infectious and acute disease such as a fever should not use this device.
* People who have hemorrhagic disease, vascular ruptures, skin inflammation, or any disease of the skin should not use this device.
* People who have immune system dysfunction such as Leukemia, Hemophilia, etc., and light sensitive persons should not use this device.
* Individuals with a history of melanoma, raised moles, suspicious lesions, keloid scar formation, or healing problems should not undergo laser light therapy.
* Individuals with active infections, open lesions, hives, herpetic lesions, cold sores, or tattoos and permanent make-up in the area of treatment should not undergo laser light therapy.
* People who have used isotretinoin (commonly known as Accutane), tetracycline, St. John's Wort, or any photo sensitizing drugs in the last year should not undergo laser light therapy.
* Individuals with autoimmune diseases such as Lupus, Scleroderma, or Vitiligo should not undergo laser light therapy.
* Individuals who have pacemakers or other electro-stimulation devices surgically implanted should not undergo laser light therapy.
* Any insulin dependent individual should consult their physician before undergoing laser light therapy.
* All individuals considered "vulnerable" such as children, pregnant women, nursing home residents or other institutionalized persons, students, employees, fetuses, prisoners, and persons with decisional incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-02-09 (Actual); Study Completion 2019-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Namynanik, BS, Study Director
Locations (1):
- Cross Chiropractic Center, Hixson, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Trial recruitment period had a start date of January 14th and ended on January 19th 2019. (A total of 6 days) All participant recruitment and interviews were conducted at the Cross Chiropractic Center in Hixson, TN.
Groups:
- Care as Usual Group: A randomly selected group of approximately 20 participants who will receive treatment per the prescribed trial protocol using a fully functional invisa-RED Technology Elite device. Treatment protocol is as follows: Participants will undergo nine (9) therapy sessions of 20 minutes each over a three week period; using a singular Low-level Laser Therapy (LLLT) protocol setting for pulse (3.5s) and delay (0.2s), however power settings will be based on the participants Fitzpatrick Scale skin type. For skin types i and ii a power setting of 7 will be used, for skin types iii and iv a power setting of 6, for skin types v and vi a power setting of 4 will be employed.
  Care as Usual Group: Each participant randomly assigned to the "Care As Usual Group" will undergo nine therapy sessions over three weeks using a fully functioning invisa-RED Technology Elite device.
- Sham Group: A randomly selected group of approximately 20 participants who will receive treatment per the prescribed trial protocol using a non functional invisa-RED Technology Elite device. (The sham device will be disabled and will deliver no Low-level Laser Light energy during therapy.) Treatment protocol is as follows: Participants will undergo nine (9) therapy sessions of 20 minutes each over a three week period; using a singular protocol setting for pulse (3.5s) and delay (0.2s), however power settings will be based on the participants Fitzpatrick Scale skin type. For skin types i and ii a power setting of 7 will be used, for skin types iii and iv a power setting of 6, for skin types v and vi a power setting of 4 will be employed.
  Sham Group: Each participant randomly assigned to the "Sham Group" will undergo nine therapy sessions over three weeks using a non functioning invisa-RED Technology Elite device.
Period: Overall Study
Arm/Group | Care as Usual Group | Sham Group
Started | 20 | 19
Completed | 18 | 15
Not Completed | 2 | 4
Not completed — Lack of Efficacy, Withdrawal by Subject | 0 | 4
Not completed — Unable to measure body fat percentage | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Care as Usual Group: A randomly selected group of 20 participants who will receive treatment per the prescribed trial protocol using a fully functional invisa-RED Technology Elite device. Treatment protocol is as follows: Participants will undergo nine (9) therapy sessions of 20 minutes each over a three week period; using a singular LLLT protocol setting for pulse (3.5s) and delay (0.2s), however power settings will be based on the participants Fitzpatrick Scale skin type. For skin types i and ii a power setting of 7 will be used, for skin types iii and iv a power setting of 6, for skin types v and vi a power setting of 4 will be employed.
  Care as Usual Group: Each participant randomly assigned to the "Care As Usual Group" will undergo nine therapy sessions over three weeks using a fully functioning invisa-RED Technology Elite device.
- Total: Total of all reporting groups
Arm/Group | Care as Usual Group | Sham Group | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (9.22) | 50.6 (13.30) | 49.46 (11.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 1 | 3 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39
Percentage Body Fat [Mean (Standard Deviation); unit: Percent Body Fat] — Body fat percentage measured using Bioelectrical Impedance Analysis (BIA) device, measurement protocol maintained strict adherence to the manufacturers directions for use. Population: 1. Number of "Care as Usual Group" participants measured was reduced by two morbidly obese participants whose body fat percentage could not be accurately measured.
  2. Number of Sham Group was reduced by a drop out of 4 participants due to schedule conflicts and lack of efficacy.
  Percent Body Fat
    number analyzed (Participants) | 18 | 15 | 33
    (all) | 40.38 (6.25) | 39.63 (6.90) | 40.04 (6.46)
Body Circumference Measurements [Mean (Standard Deviation); unit: Inches] — Prior to the initial therapy session body measurements are made of each participants' chest, right arm, upper-waist, mid-waist, hips, and right thigh, they are then summed and the total recorded. Population: Number of Sham Group was reduced by a drop out of 4 participants due to schedule conflicts and lack of efficacy.
  Inches
    number analyzed (Participants) | 20 | 15 | 35
    (all) | 225.19 (30.64) | 222.58 (24.83) | 224.07 (27.93)
Weight of Body Fat [Mean (Standard Deviation); unit: Pounds] — In order to measure each participants body fat in pounds, the percentage of body fat for each participant was measured prior to the start of any therapy using Bioelectrical Impedance Analysis (BIA). The percentage is then multiplied by the total body weight of the participant in order to compute the weight in pounds of the participants body fat. Population: 1. Number of "Care as Usual Group" participants measured was reduced by two morbidly obese participants whose body fat percentage could not be accurately measured.
  2. Number of Sham Group was reduced by a drop out of 4 participants due to schedule conflicts and lack of efficacy.
  Pounds
    number analyzed (Participants) | 18 | 15 | 33
    (all) | 82.80 (28.12) | 85.81 (26.06) | 84.17 (26.83)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Fat Percentage
Description: Measured change in body fat as a percentage of total weight.
Time Frame: In order to determine change over time, body fat as a percentage of body weight will be measured before any treatment at first therapy session and measured again for comparison at the end of three weeks therapy.
Population: 1. Number of "Care as Usual Group" participants measured was reduced by two morbidly obese participants whose body fat percentage could not be accurately measured.
  2. Number of Sham Group was reduced by a drop out of 4 participants due to schedule conflicts and lack of efficacy.
Measure: Mean (95% Confidence Interval); unit: Percentage of Body Fat
Groups:
- Care as Usual Group: A randomly selected group of approximately 20 participants who will receive treatment per the prescribed trial protocol using a fully functional invisa-RED Technology Elite device. Treatment protocol is as follows: Participants will undergo nine (9) therapy sessions of 20 minutes each over a three week period; using a singular LLLT protocol setting for pulse (3.5s) and delay (0.2s), however power settings will be based on the participants Fitzpatrick Scale skin type. For skin types i and ii a power setting of 7 will be used, for skin types iii and iv a power setting of 6, for skin types v and vi a power setting of 4 will be employed.
  Care as Usual Group: Each participant randomly assigned to the "Care As Usual Group" will undergo nine therapy sessions over three weeks using a fully functioning invisa-RED Technology Elite device.
- Sham Group: A randomly selected group of approximately 20 participants who will receive treatment per the prescribed trial protocol using a non functional invisa-RED Technology Elite device. (The sham device will be disabled and will deliver no low laser light energy during therapy.) Treatment protocol is as follows: Participants will undergo nine (9) therapy sessions of 20 minutes each over a three week period; using a singular protocol setting for pulse (3.5s) and delay (0.2s), however power settings will be based on the participants Fitzpatrick Scale skin type. For skin types i and ii a power setting of 7 will be used, for skin types iii and iv a power setting of 6, for skin types v and vi a power setting of 4 will be employed.
  Sham Group: Each participant randomly assigned to the "Sham Group" will undergo nine therapy sessions over three weeks using a non functioning invisa-RED Technology Elite device.
Arm/Group | Care as Usual Group | Sham Group
Number analyzed (Participants) | 18 | 15
Percentage of Body Fat | -1.7556 [-2.4273 to -1.0838] | 0.280 [-.1194 to 0.6794]
Statistical Analysis 1: Comparison: Care as Usual Group vs Sham Group; The null hypothesis states that in the population from where the sample was obtained there was no difference between the intervention (invisa-RED Elite) and placebo groups in the mean change in the primary outcome variable, i.e. Change in Body Fat Percentage; Test type: Superiority; p < 0.01, t-test, 2 sided — p-value is calculated using SPSS; Mean Difference (Net) = 2.036, 95% CI 2-sided [1.243 to 2.828]
Statistical Analysis 2: Comparison: Care as Usual Group vs Sham Group; A single sample Kolmogorov-Smirnov normality test was used to examine if variables are normally distributed for the population from which the trial groups are drawn. The null hypothesis is that the distribution of Percent of Body Fat Lost or Gained is normal with mean -.83 and standard deviation 1.50218; Test type: Other; p = 0.20, Kolmogorov-Smirnov Test — The significance value has been Lilliefors corrected and represents the lower bound of the true significance
Statistical Analysis 3: Comparison: Care as Usual Group vs Sham Group; To test that the trial participant's population variances are equal (or exhibit homogeneity of variance), a Levene's Test for Equality of Variance was conducted. It tests the null hypothesis that the population variances are equal (called homogeneity of variance or homoscedasticity). For this test if the resulting p-value of Levene's test is less than .05, the obtained differences in sample variances are unlikely to have occurred based on random sampling from a population with equal variances; Test type: Other; p = 0.075, Levene's Test for Equality of Variance

2. Primary Outcome: Change in Body Circumference Measurements
Description: The prescribed body circumference measurements of the chest, right arm, upper-waist, mid-waist, hips, and right thigh are summed for each participant and recorded.
Time Frame: In order to determine change over time, the prescribed body measurements will be summed for each participant and recorded before any treatment at first therapy session and recorded again for comparison at the end of three weeks therapy.
Population: Number of Sham Group was reduced by a drop out of 4 participants due to schedule conflicts and lack of efficacy.
Measure: Mean (95% Confidence Interval); unit: Inches
Arm/Group | Care as Usual Group | Sham Group
Number analyzed (Participants) | 20 | 15
Inches | -10.162500 [-12.1930 to -8.1319] | -3.100000 [-5.8958 to -.304128]
Statistical Analysis 1: Comparison: Care as Usual Group vs Sham Group; Designed as a superiority trial with the aim of establishing whether the intervention was superior or inferior to a placebo in effectiveness as a therapy for change over time in measured body circumference. The null hypothesis states that in the population from where the sample was obtained there was no difference between the intervention (invisa-RED Elite) and placebo groups in the mean change in the primary outcome variable, i.e. measured body circumference; Test type: Superiority; p < 0.01, t-test, 2 sided — p-value is calculated using SPSS; Mean Difference (Net) = 7.063, 95% CI 2-sided [3.829 to 10.296]
Statistical Analysis 2: Comparison: Care as Usual Group vs Sham Group; A Kolmogorov-Smirnov normality test was used to examine if variables are normally distributed for the population from which the trial groups are drawn. The null hypothesis is that the distribution of Total Inches Lost or Gained is normal with mean -7.136 and standard deviation 5.796; Test type: Other; p = 0.20, Kolmogorov-Smirnov Test — The significance value has been Lilliefors corrected and represents the lower bound of the true significance
Statistical Analysis 3: Comparison: Care as Usual Group vs Sham Group; [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.44, Levene's Test for Equality of Variance

3. Primary Outcome: Change in Weight of Body Fat
Description: The percentage of body fat for each participant was measured using Bioelectrical Impedance Analysis (BIA). That percentage is then multiplied by the total body weight of the participant in order to calculate the weight in pounds of the participants body fat.
Time Frame: In order to determine change over time, each participants body fat weight will be calculated before any treatment at the first therapy session and calculated again to determine if there exists any change at the end of three weeks therapy.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Care as Usual Group | Sham Group
Number analyzed (Participants) | 18 | 15
Pounds | -4.5183 (3.42558) | -.0480 (2.35970)
Statistical Analysis 1: Comparison: Care as Usual Group vs Sham Group; Designed as a superiority trial with the aim of establishing whether the intervention was superior or inferior to a placebo in effectiveness as a therapy for change in body fat, measured in pounds. The null hypothesis states that in the population from where the sample was obtained there was no difference between the intervention (invisa-RED Elite) and placebo groups in the mean change in the primary outcome variable, i.e. change in pounds of body fat; Test type: Superiority; p < 0.01, t-test, 2 sided — p-value is computed using SPSS; Mean Difference (Net) = 4.4703, 95% CI 2-sided [2.3372 to 6.6034]
Statistical Analysis 2: Comparison: Care as Usual Group vs Sham Group; A single sample Kolmogorov-Smirnov normality test was used to examine if variables are normally distributed for the population from which the trial groups are drawn. The null hypothesis is that the distribution of the Weight of Body Fat Lost or Gained is normal with mean -2.49 and standard deviation 3.71209; Test type: Other; p = .200, Kolmogorov-Smirnov Test — The significance value has been Lilliefors corrected and represents the lower bound of the true significance
Statistical Analysis 3: Comparison: Care as Usual Group vs Sham Group; [analysis description as in outcome 1, analysis 3]; Test type: Other; p = .438, Levene's Test for Equality of Variance

ADVERSE EVENTS:
Time Frame: Three weeks concurrent with clinical trial.
Description: Participants were instructed to immediately notify the attending clinician during each therapy session if they experienced any discomfort. Clinicians were trained to recognize any adverse effects such as extreme skin redness or blistering and instructed to report any such occurrence.
Arm/Group | Care as Usual Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/15
Other Adverse Events (participants affected / at risk) | 0/20 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT03811093/Prot_001.pdf
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT03811093/SAP_000.pdf